CLINICAL TRIAL: NCT04403334
Title: Postoperative Safety Outcomes in Patients Undergoing Routine Phacoemulsification Cataract Surgery With Intraoperative Intracameral Injection of Preservative-Free Moxifloxacin Versus Levofloxacin
Brief Title: Postoperative Safety Outcomes of Intraoperative Intracameral Preservative-Free Moxifloxacin Versus Levofloxacin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peregrine Eye and Laser Institute (Other)
Responsible Party: Principal Investigator, Harvey Siy Uy, Medical Director, Peregrine Eye and Laser Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20180101
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Cataract Senile; Endophthalmitis; Antibiotic Side Effect; Safety Issues
Keywords: levofloxacin; moxifloxacin; prophylaxis; endophthalmitis; cataract surgery
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: unlabelled syringe containing interventional drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracameral levofloxacin (Experimental): 0.5% unpreserved solution
  Interventions: Drug: Levofloxacin Ophthalmic
- Intracameral moxifloxacin (Experimental): 0.5% unpreserved solution
  Interventions: Drug: Moxifloxacin Ophthalmic

INTERVENTIONS:
Drug: Levofloxacin Ophthalmic — 0.1 ml of unpreserved 0.5% levofloxacin
  Arms: Intracameral levofloxacin
Drug: Moxifloxacin Ophthalmic — 0.1 ml of unpreserved 0.5% moxifloxacin
  Arms: Intracameral moxifloxacin

SUMMARY:
Comparative safety study of intracameral levofloxacin versus moxifloxacin for postoperative infection prophylaxis

DETAILED DESCRIPTION:
Randomized clinical trial comparing corneal and retinal changes after intracameral levofloxacin or moxifloxacin administered at the end of surgery among eyes undergoing uncomplicated phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* Eyes undergoing uncomplicated cataract surgery by phacoemulsification

Exclusion Criteria:

* Corneal opacities, corneal dystrophies, glaucoma, uveitis, retinopathy, optic neuropathy, concomitant infection (blepharitis, hordeolum, or conjunctivitis) or uncontrolled systemic disease and intraoperative complications that may affect visual outcomes were excluded from the study

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
Endothelial Cell Count | 3 months
  Change in endothelial cell count as measured by specular microscopy
Central Retina Thickness | 3 months
  Change in central retinal thickness as measured by spectral domain optical coherence tomography

SECONDARY OUTCOMES:
Adverse Events | 3 months
  Onset of Adverse events following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Harvey S Uy, MD, Principal Investigator — Peregrine Eye and Laser Institute
Locations (1):
- Peregrine Eye and Laser Instittute, Makati City, MM, Philippines